CLINICAL TRIAL: NCT06821854
Title: A Post-market, Monocentric, Interventional, Single-arm, Confirmative Clinical Investigation to Evaluate the Performance and the Safety of PN20 (Plinest) for the Improvement of Skin Hydration
Brief Title: Efficacy and Safety of PN20 (Plinest) for the Improvement of Skin Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-PN20-2024
Record Dates: First submitted 2025-01-30; First posted 2025-02-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Skin Hydration; Skin Elasticity
Keywords: skin hydration; Polynucloetides; PN HPT; Mastelli; Plinest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: PN20 (Plinest)

INTERVENTIONS:
Device: PN20 (Plinest) — PN20 (Plinest) is a single-use viscoelastic, and sterile gel for intradermal use. PN20 contains polynucleotides (20 mg/ml- 2%), water, sodium chloride, sodium phosphate and disodium phosphate.
  PN20 is administered using a fine needle (usually 30 G) by injecting the solution into the dermis. Depending on the medical assessment, different injection techniques, such as linear threading, serial punctures, crosslinked, radial fanning or mixed, can be used. The injection site must consist of healthy skin. PN20 can also be administered by means of modern non-invasive techniques (electroporation, hydroelectrophoresis, etc.). In all these cases, thoroughly cleanse and disinfect the area to be treated before application.
  PN20, thanks to its versatility and manageability, can be used in any skin area; in the current clinical investigation the face, neck or décolleté will be treated.

SUMMARY:
This is a post-market, monocentric, interventional, single-arm, confirmative clinical investigation to evaluate the performance and the safety of PN20 (PLINEST) for the improvement of skin hydration.

Each Subject, after signing the Informed Consent Form (ICF), will enter into a screening/baseline phase during which the baseline tests will be conducted. The Subject can be treated immediately after signing the ICF.

For each Subject, 5 visits will be planned during which several assessments will be performed as described in the Flowchart:

* V0 (Screening/baseline): Day 0, when the first IP injection will be performed;
* V1: 2 weeks ± 7 days from V0, when the second IP injection will be performed;
* V2: 2 weeks ± 7 days from V1, when the third IP injection will be performed (End Of Treatment/EOT);
* V3: maximum 4 months from V0 and 2 months after the last IP injection (V2);
* V4: maximum 6 months form V0 and 4 months after the last IP injection (V2).

At V0, the Investigator will collect demographic data (e.g., gender, age, skin phototype according to Fitzpatrick's classification), medical history (e.g., history of autoimmune disease, diabetes, etc.), drug allergy history of the enrolled Subject.

At V0, V1, and V2 according to the instructions for use (IFU), the enrolled Subjects will be treated with PN20 in maximum 2 areas of the face, or 1 area of the face plus neck/décolleté, making sure that at least 14 areas for face, neck and décolleté will be reached.

Local anesthetics containing lidocaine may be used in order to guarantee the necessary comfort to the Subject.

Performance will be evaluated by the Investigator using the Global Aesthetic Improvement Scale (GAIS) at each visit. The GAIS will be independently completed by the Investigator and the Subject. Photographs with a 2D camera will be taken at each visit. Skin hydration will be assessed by using the MoistureMeterEpiD (at least three measurements will be obtained per each area treated) at each visit.

Skin elasticity will be evaluated using the ElastiMeter (at least three measurements will be obtained per each area treated) at each visit.

Skin turgor will be assessed by the Investigator using a 5-Likert scale at each visit.

At V0, V1 and V2 after injection, the Investigator will record Subjects' pain intensity using the Numerical Rating Scale (NRS).

Subject satisfaction with treatment will be evaluated with a 5-point Likert Scale at V3 and EOS visit (V4).

Safety will include evaluation of possible cutaneous reactions at each visit. Adverse events, concomitant medications, and device deficiencies will be monitored during the entire duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject Informed consent form (ICF) signed;
2. Female and male Subjects aged 18-70 years;
3. Subjects desiring improvement of skin hydration in maximum 2 areas of the face, or 1 area of the face plus neck or décolleté;
4. Healthy skin;
5. Willingness to discontinue all dermatological treatment and procedures during the study;
6. Willingness to follow all study procedures, including attending all site visits, tests and examinations;
7. Agreeing to present at each study visit without face/neck/ décolleté cosmetics;
8. Accepting to not change their habits regarding food, physical activity, face/neck/décolleté cosmetics and cleansing products;
9. Willingness to follow indications to minimize exposure of the treated area to too much sunlight or extreme cold, at least until the papules have completely subsided;
10. Skin phototype I-IV according to Fitzpatrick's classification.

Exclusion Criteria:

1. Other - different - clinical conditions of the skin (i.e. rosacea, psoriasis, vitiligo, active eczema, severe scleroderma, severe acne and diagnosticated cancer with/without ongoing antitumor therapy);
2. Infectious or inflammatory processes near the area of intervention;
3. Presence of cutaneous disease on the tested area, as malformations and recurrent facial/labial herpes;
4. Presence of tendon, bone or muscular implants near the area of intervention;
5. Ongoing cutaneous allergies;
6. Allergy or contraindications to device components;
7. Concomitant intake of anticoagulant or antiplatelet medications;
8. Subjects who have not followed a washout period of 2 weeks from topical corticosteroids, antibiotics, benzoyl-peroxide, azelaic acid, hydroxy acids, topical retinoids;
9. Immune system illnesses/disease;
10. Uncontrolled diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder);
11. Treatment with substances which act on blood fluidity (eg. Aspirin, NSAIDs, Vitamin E), or drugs able to influence the test results in the investigator opinion, within 5 days prior to study inclusion;
12. Known drug and/or alcohol abuse;
13. Mental incapacity that precludes adequate understanding or cooperation;
14. Any previous permanent and non-permanent cutaneous treatment for aesthetic correction (biomaterial implant, lifting, laser, botulinum toxin injections, chemical peeling, fillers) of the treated area within 6 months prior to study inclusion;
15. Pregnancy or breastfeeding;
16. Participation in another investigational study within 1 month prior to study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Global Aesthetic Improvement Scale (GAIS) from V4 to baseline completed by Investigator | From enrollment to the end after 4 months from the last treatment.
  To evaluate the performance of PN20 on the aesthetic appearance of the skin 4 months after the last treatment, the change in the Global Aesthetic Improvement Scale (GAIS), rated on a 5-point scale (1= very much/extremely improved; 2= much improved; 3= improved; 4= no change; 5= worse) from V4 to baseline (pre-treatment), will be assessed. The GAIS will be completed by the Investigator.
  The pre-treatment GAIS score (at baseline/V0) will be "4" for each treated area for all enrolled subjects.

SECONDARY OUTCOMES:
Change in Investigator and Subject Global Aesthetic Improvement Scale (GAIS) at each visit | From enrollment to the end after 4 months from the last treatment (at each visit)
  To evaluate the performance of PN20 on the aesthetic appearance of the skin, the change in the Global Aesthetic Improvement Scale (GAIS), rated on a 5-point scale (1= very much/extremely improved; 2= much improved; 3= improved; 4= no change; 5= worse), will be assessed at each visit. The GAIS will be completed independently by the Investigator and the Subject.
Performance of PN20 on the skin hydration at each visit | From enrollment to the end after 4 months from the last treatment (at each visit)
  To evaluate the performance of PN20 on skin hydration at each visit, the MoistureMeterEpiD, which displays percentage water content (0 - 100 %), will be used by the Investigator.
Performance of PN20 on skin elasticity at each visit | From enrollment to the end after 4 months from the last treatment (at each visit)
  To evaluate the performance of PN20 on skin elasticity at each visit, the ElastiMeter, which measures skin elasticity in N/m, will be used by the Investigator at each visit.
Performance of PN20 on skin turgor at each visit | From enrollment to the end after 4 months from the last treatment (at each visit)
  To evaluate the performance of PN20 on skin turgor at each visit, a 5-Likert scale (1 - Very poor, 2 - Poor, 3 - Good, 4 - Very good, 5 - Excellent) will be used by the Investigator at each visit.
Pain intensity after injection of PN20 | Visit 0 (Baseline), Visit 1 and Visit 2
  To evaluate pain intensity after injection of PN20, a Numerical Rating Scale (NRS), a 0 to 10 scale indicating the degree of pain the patient experienced (0 - No Pain, 5 - Moderate Pain, 10 - Worst possible Pain), will be used at Visit 0 (Baseline), Visit 1 and Visit 2.
Subject satisfaction with PN20 | Visit 3 and at End of study (Visit 4)
  To evaluate subject satisfaction with PN20, a 5-Likert scale, from 1 to 5 indicating how satisfied is the patient (1 - Extremely dissatisfied, 5 - Extremely satisfied), will be used at Visit 3 and at End of study (Visit 4)
Device deficiencies | Baseline (Visit 0), Visit 1, and Visit 2
  A device deficiency (DD) is any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in information supplied by the manufacturer.
  This definition includes device deficiencies related to the investigational medical device.
  The rate of DD will be assessed and counted by the investigator at baseline (Visit 0), at Visit 1 and at Visit 2.
Adverse events, serious adverse events and concomitant medications monitoring | All visits from baseline to the last follow-up after 12 weeks from the end of the treatment
  Adverse events, serious adverse events and concomitant medications will be monitored during the entire study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica di Chirurgia plastica e ricostruttiva/Ospedale Policlinico San Martino, Genova, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] E. Bartoletti et al., "PN HPTTM and Striae Albae-Exploratory Interim Analysis of a Randomised Prospective Study," Surgical Research, vol. 5, no. 3, Sep. 2023, doi: 10.33425/2689-1093.1057
- [Background] Lim TS, Liew S, Tee XJ, Chong I, Lo FJ, Ho MJ, Ong K, Cavallini M. Polynucleotides HPT for Asian Skin Regeneration and Rejuvenation. Clin Cosmet Investig Dermatol. 2024 Feb 13;17:417-431. doi: 10.2147/CCID.S437942. eCollection 2024. PMID 38371328
- [Background] Araco A, Araco F. Preliminary Prospective and Randomized Study of Highly Purified Polynucleotide vs Placebo in Treatment of Moderate to Severe Acne Scars. Aesthet Surg J. 2021 Jun 14;41(7):NP866-NP874. doi: 10.1093/asj/sjab125. PMID 33755110
- [Background] De Caridi G, Massara M, Acri I, Zavettieri S, Grande R, Butrico L, de Franciscis S, Serra R. Trophic effects of polynucleotides and hyaluronic acid in the healing of venous ulcers of the lower limbs: a clinical study. Int Wound J. 2016 Oct;13(5):754-8. doi: 10.1111/iwj.12368. Epub 2014 Sep 16. PMID 25224018
- [Background] Cavallini M, Bartoletti E, Maioli L, Massirone A, Pia Palmieri I, Papagni M, Priori M, Trocchi G; As Members of The Polynucleotides HPT Priming Board, Collegio Italiano delle Societa Scientifiche di Medicina Estetica (Italian College of the Aesthetic Medicine Scientific Societies) - SIME, AGORA, SIES. Consensus report on the use of PN-HPT (polynucleotides highly purified technology) in aesthetic medicine. J Cosmet Dermatol. 2021 Mar;20(3):922-928. doi: 10.1111/jocd.13679. Epub 2020 Sep 21. PMID 32799391